CLINICAL TRIAL: NCT05542576
Title: Prospective Randomized Open, Blinded Endpoint (PROBE) Study of AMDX-2011P as a Retinal Tracer in Subjects With Neurodegenerative Diseases Associated With Amyloidogenic Proteinopathy
Brief Title: Study of AMDX-2011P as a Retinal Tracer in Subjects With Neurodegenerative Diseases Associated With Amyloidogenic Proteinopathy
Acronym: PROBE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amydis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: AMDX-2011P-101
Record Dates: First submitted 2022-09-07; First posted 2022-09-15 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease; Amyotrophic Lateral Sclerosis
Keywords: Parkinsons; ALS
MeSH Terms: conditions — Parkinson Disease; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Dose escalating via Cohorts total 1-3 cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AMDX2011P 25mg (Experimental): 25mg (1ml) single bolus injection intravenous for diagnostic review
  Interventions: Drug: AMDX2011P
- AMDX2011P 50mg (Experimental): AMDX2011P 50mg (2ml) single bolus injection intravenous for diagnostic review
  Interventions: Drug: AMDX2011P
- AMDX2011P 100mg (Experimental): AMDX2011P 100mg (4ml) single bolus injection intravenous for diagnostic review
  Interventions: Drug: AMDX2011P

INTERVENTIONS:
Drug: AMDX2011P — AMDX2011P single bolus injection intravenous for diagnostic review

SUMMARY:
The purpose of this research study is to assess safety and tolerability of a single intravenous (given through a vein) dose of the investigational retinal tracer AMDX-2011P in patients with neurodegenerative diseases (Parkinson's disease and ALS).

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of three different doses of AMDX-2011P (25mg, 50mg, or 100mg) given as a single intravenous dose in patients with neurodegenerative diseases (Parkinson's disease and ALS). The first cohort of participants taking part in the study will receive the lowest dose of AMDX-2011P (25mg). If no major side effects occur, the dose will be increased for the next group of participants to 50mg and then to 100mg.

Secondary objective of this study is to characterize the pharmacokinetic (PK) profile of AMDX-2011P and AMDX-2011.

Exploratory evaluations of the biological activity of AMDX-2011P in the retina will be performed by imaging.

ELIGIBILITY:
Inclusion Criteria:

For Subjects with Parkinson's Disease

1. Clinically established Parkinson's disease based on Movement Disorder Society (MDS) Clinical Diagnostic Criteria for Parkinson's disease (Table 8) and a modified Hoehn & Yahr scale of 1-3 (Table 9).
2. No suspected atypical parkinsonian syndromes due to drugs, metabolic disorders, encephalitis, or degenerative diseases.

   For Subjects with ALS
3. Confirmed diagnosis of ALS with both upper and lower motor neuron involvement.

   For All Subjects
4. Ability to undergo retinal imaging.
5. Subject or legally authorized representative must provide signed informed consent (or signed assent form) prior to study entry and have the ability and willingness to attend and comply with the necessary study procedures and visits at the study site. For subjects unable to physically sign the informed consent, a guardian or trusted care giver can sign on their behalf in presence of an independent witness.
6. Contraception use by study subjects of childbearing potential (male and female) and female partners of childrearing potential male subjects should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

1. Presence of any underlying physical or psychological medical condition that would make it unlikely that the subject will complete the study per protocol.
2. Clinically significant laboratory abnormalities assessed by the investigator.
3. Active malignancy and/or history of malignancy in the past 5 years, with the exception of completely excised non-melanoma skin cancer or low-grade cervical intraepithelial neoplasia.
4. Prolonged QTcF (>450 ms for males and >470 ms for females), cardiac arrhythmia, or any clinically significant abnormality in the resting ECG, as judged by the investigator.
5. Presence of any ocular condition that would significantly hinder the ability to detect and quantify hyper-fluorescent puncta (e.g., eyes with significant hyper-autofluorescence that would mask the ability to detect, quantify, and discern post-injection hyper-fluorescent signal from pre-injection hyper-autofluorescence signal).
6. Use of any new prescription therapies or vaccines within 7 days prior to the study drug administration.
7. Drugs with potential phototoxicity per Package Insert are prohibited within 48 hours or 5 half-lives, whichever is longer, prior to first study drug until End-of-study (EOS) visit, except for those required for treatment of underlying disease.
8. Administration of investigational product in another study within 30 days prior to the first study drug administration, or five half-lives, whichever is longer.
9. Females who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masoud Mokhtarani, MD, Study Chair — Amydis Inc.
Locations (2):
- United States (2):
  - Eye Research Foundation, Newport Beach, California
  - Brittany NIcholl, Pasadena, California

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data at this time.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 13 subjects: 3 in Cohort 1 (25mg dose) 4 in Cohort 2 (50mg dose) 6 in Cohort 3 (100mg dose)
Groups:
- AMDX2011P 25mg: AMDX2011P 25mg (1ml) single bolus injection intravenous for diagnostic review
Period: Overall Study
Arm/Group | AMDX2011P 25mg | AMDX2011P 50mg | AMDX2011P 100mg
Started | 3 | 4 | 6
Completed | 3 | 4 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AMDX2011P 25mg | AMDX2011P 50mg | AMDX2011P 100mg | Total
Number analyzed (Participants) | 3 | 4 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 2 | 5
  >=65 years | 2 | 2 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 0 | 4
  Male | 2 | 1 | 6 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 4 | 6 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: AMDX-2011P Adverse Events Profile
Description: Incidence of Treatment Emergent Adverse Events (TEAEs) at for each cohort (dose level).
Time Frame: 1 week
Measure: Number; unit: Treatment Emergent Adverse Events TEAEs
Arm/Group | AMDX2011P 25mg | AMDX2011P 50mg | AMDX2011P 100mg
Number analyzed (Participants) | 3 | 4 | 6
Treatment Emergent Adverse Events TEAEs | 0 | 1 | 3

2. Secondary Outcome: Concentration of AMDX-2011P
Description: Peak Plasma Concentration (Cmax)
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AMDX2011P 25mg | AMDX2011P 50mg | AMDX2011P 100mg
Number analyzed (Participants) | 3 | 3 | 6
ng/mL | 4400 (572) | 16600 (15800) | 14600 (3890)

3. Secondary Outcome: Pharmacokinetic Analysis of AMDX-2011P
Description: Area under the plasma concentration versus time curve (AUC)
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | AMDX2011P 25mg | AMDX2011P 50mg | AMDX2011P 100mg
Number analyzed (Participants) | 3 | 3 | 6
h*ng/mL | 706 (110) | 3170 (3290) | 2330 (637)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 8 days
Arm/Group | AMDX2011P 25mg | AMDX2011P 50mg | AMDX2011P 100mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 0/3 | 1/4 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMDX2011P 25mg (N=3) | AMDX2011P 50mg (N=4) | AMDX2011P 100mg (N=6)
Altered taste (Nervous system disorders) | 0 | 1 | 1 — Mild
Paresthesia (Nervous system disorders) | 0 | 0 | 2 — Mild
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 — Mild
Anxiety (Psychiatric disorders) | 0 | 1 | 0 — Mild
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 — Mild
Feeling Hot (General disorders) | 0 | 0 | 1 — Mild

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT05542576/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/76/NCT05542576/SAP_001.pdf